CLINICAL TRIAL: NCT05123898
Title: Comparative Analysis of the Effectiveness of Free Connective Tissue Graft and Xenogenic Collagen Matrix Transplantation in Patients With Dental Implants.
Brief Title: Clinical and Histological Outcomes of Using Collagen Matrix or Soft Tissue Graft Around Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09102019
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Soft Tissue Atrophy
Keywords: connective tissue graft; xenogeic collagen matrix; increasing of soft tissue thickness; dental implant; soft tissue augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 group (Other): The patients underwent implant placement in combination with an increase in the thickness of soft tissues using a free connective tissue graft from the tuber region on the upper jaw.
  Interventions: Procedure: Soft tissue augmentation
- 2 group (Experimental): The patients underwent implant placement in combination with an increase in the thickness of soft tissues using collagen matrix "Fibromatrix"
  Interventions: Procedure: Soft tissue augmentation

INTERVENTIONS:
Procedure: Soft tissue augmentation — 1. Incision the mucosa at the alveolar ridge, mucosal-periosteal flap elevation
  2. Placement of the Ostem dental implant (Osstem Implant Co., Ltd.)
  3. Modeling of sterile collagen matrix according to the shape of the recipient bed
  4. Fixation of the collagen matrix to the vestibular flap
  5. Suturing the wound tightly

SUMMARY:
This was an interventional prospective randomized clinical trial (RCT) in parallel groups. The sample size is 35 patients who were randomly divided into two groups depending on the surgical intervention used. First group - patients underwent increasing the thickness of the mucous membrane using free connective tissue graft from tuberosity area of the upper jaw. Second group - patients used collagen matrix "Fibromatrix" (LLC "Cardioplant", Russia; registration in Russia 20/05/2019 No FSZ 2019/83671). In the postoperative period the value of soft tissue thickness gain, duration of surgery, severity of pain syndrome and quality of life were assessed. Also, after 3 months simultaneously with installation of gingiva formers biopsy specimens were sampled with mucotome in the area of the intervention followed by histomorphometric analysis of the obtained biopsies.

DETAILED DESCRIPTION:
The aim of this research was to perform a comparative clinical and histomorphometric analysis of soft tissues in the area of soft tissue graft and collagen matrix transplantation. Thirty five patients diagnosed with partial absence of teeth were examined on the basis of the Department of Surgical Dentistry of the E.V. Borovsky Institute of Dentistry of I.M. Sechenov First Moscow State Medical University. Patients had a soft tissue thickness deficiency from the vestibular surface in the area of the planned dental implant placement which was an indication for its increase. All patients were randomly divided into two groups depending on method of soft tissue augmentation used. In 1 group (n=15) transplantation of a free connective tissue graft (CTG) from tuberosity area of the upper jaw was performed. In 2 group (n=20) collagen matrix "Fibromatrix" was used. According to gender and age characteristics both groups were comparable. Randomization of patients was carried out at the stage of surgical intervention as follows: after a dental implant placement and preparation of recipient's bed an envelope with a randomly assigned treatment method (using a connective tissue graft or a collagen matrix) was opened.

During the operation, incision was made along the top of the alveolar ridge within the defect; a full-thickness muco-periosteal flap was elevated. Traditional 2-stage dental implantation was performed according to surgical protocols of dental implant systems Ostem (Osstem Implant Co., Ltd., Korea; registration in Russia 05.09.2018 No FSZ 2018/7577). A free connective tissue graft was harvested in patients of the first group. Graft was fixed with a horizontal U-shaped suture to the buccal muco-periosteal flap. In second patients group a fragment of the collagen matrix "Fibromatrix" was fixed to the buccal muco-periosteal flap (LLC "Cardioplant", Russia; registration in Russia 20.05.2019 No № FSZ 2019/83671). For patients of all groups mobilization of the muco-periosteal flap conducted followed by suturing the wound tightly without tension with simple interrupted sutures.

In the early postoperative period the standard antibacterial and anti-inflammatory therapy in combination with the use of local antiseptics for daily care was prescribed. The stage of the implant uncovering with hilling abutments installation was carried out 3 months after the intervention. At this stage, a soft tissue fragment was taken using a mucotome in the area of the previously performed mucous membrane thickness increasing for subsequent histomorphometric analysis. In the study we used both conventional light microscopy (microscopy in the light field) and polarizing microscopy - to estimate the content of collagen fibers in preparations stained with picrosirius red. During a morphometric study we carried out a quantitative assessment of the characteristics of the epithelial layer, the basement membrane relative length (the ratio of the absolute length of the basement membrane to the length of the epithelial layer), the characteristics of the underlying connective tissue.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of written informed consent of the patient to participate in the study;
2. The presence of an included defect (1 teeth) in the distal part of the lower jaw with a sufficient volume of bone tissue;
3. Deficiency of soft tissue thickness;
4. Adjacent teeth are without any of periodontal disease, namely the absence of periodontal probing depth > 3 mm in any site of adjacent teeth;

6. Satisfactory level of oral hygiene, namely full mouth plaque score < 20% and full mouth bleeding score < 20%;

Non-inclusion criteria:

1. The presence of concomitant pathology in the stage of decompensation;
2. Hard smokers (more than 10 cigarettes per day);
3. Radio and chemotherapy in history over the past 5 years;
4. Pregnancy and breastfeeding;
5. Taking medications that affect the healing of soft tissues (nonsteroidal anti-inflammatory drug, steroid drugs).

Exclusion Criteria:

1. Patients with infections either periodontally or periapically;
2. Pregnantcy following entrance into the study;
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures;
4. Subjects, who in the opinion of the investigator, for any reason will not be able to complete the study per protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
The amount of soft tissue thickness gain | Days 90
  To carry out the measurement an optical impression will be taken using the Primescan intraoral scanner (Dentsply/SIRONA) before the operation and on the 90th day after the operation. Further, in the specialized program GOM Inspect the stl-files will be compared and the vestibular contour changes will be evaluated at 3 equidistant points in the coronary-apical direction.

SECONDARY OUTCOMES:
VAS scale | 1 day
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
VAS scale | 3 days
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
VAS scale | 5 days
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
VAS scale | 7 days
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
VAS scale | 30 days
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
VAS scale | 90 days
  Evaluation of the severity of pain syndrome is carried out after surgery using a questionnaire, where : 0 - absence of pain; 1-2 - weak pain; 2-3 - moderate pain; 4-5 - moderate-severe pain; 6-7 - severe pain; 8-10 - unbearable pain.
OHIP-14 questionnaire | 0 day
  Description: Evaluation of the patients' quality of life is carried out using a questionnaire. Depending on the severity of the trait it is necessary to answer the following questions from 0 to 4 points: Have you had trouble pronouncing any words because of problems with your teeth or mouth? Have you felt that your sense of taste has worsened because of problems with your teeth or mouth? Have you had painful aching in your mouth? Have you found it uncomfortable to eat any foods because of problems with your teeth or mouth? Have you been self-conscious because of your teeth or mouth? Have you felt tense because of problems with your teeth or mouth? Has been your diet been unsatisfactory because of problems with your teeth of mouth? Have you had to interrupt meals because of problems with your teeth or mouth? Have you found it difficult to relax because of problems with your teeth or mouth? Have you been a bit embarrassed because of problems with your teeth or mouth? Have you been a bit
OHIP-14 questionnaire | 7 days
  Description: Evaluation of the patients' quality of life is carried out using a questionnaire. Depending on the severity of the trait it is necessary to answer the following questions from 0 to 4 points: Have you had trouble pronouncing any words because of problems with your teeth or mouth? Have you felt that your sense of taste has worsened because of problems with your teeth or mouth? Have you had painful aching in your mouth? Have you found it uncomfortable to eat any foods because of problems with your teeth or mouth? Have you been self-conscious because of your teeth or mouth? Have you felt tense because of problems with your teeth or mouth? Has been your diet been unsatisfactory because of problems with your teeth of mouth? Have you had to interrupt meals because of problems with your teeth or mouth? Have you found it difficult to relax because of problems with your teeth or mouth? Have you been a bit embarrassed because of problems with your teeth or mouth? Have you been a bit
OHIP-14 questionnaire | 30 days
  Description: Evaluation of the patients' quality of life is carried out using a questionnaire. Depending on the severity of the trait it is necessary to answer the following questions from 0 to 4 points: Have you had trouble pronouncing any words because of problems with your teeth or mouth? Have you felt that your sense of taste has worsened because of problems with your teeth or mouth? Have you had painful aching in your mouth? Have you found it uncomfortable to eat any foods because of problems with your teeth or mouth? Have you been self-conscious because of your teeth or mouth? Have you felt tense because of problems with your teeth or mouth? Has been your diet been unsatisfactory because of problems with your teeth of mouth? Have you had to interrupt meals because of problems with your teeth or mouth? Have you found it difficult to relax because of problems with your teeth or mouth? Have you been a bit embarrassed because of problems with your teeth or mouth? Have you been a bit
OHIP-14 questionnaire | 90 days
  Description: Evaluation of the patients' quality of life is carried out using a questionnaire. Depending on the severity of the trait it is necessary to answer the following questions from 0 to 4 points: Have you had trouble pronouncing any words because of problems with your teeth or mouth? Have you felt that your sense of taste has worsened because of problems with your teeth or mouth? Have you had painful aching in your mouth? Have you found it uncomfortable to eat any foods because of problems with your teeth or mouth? Have you been self-conscious because of your teeth or mouth? Have you felt tense because of problems with your teeth or mouth? Has been your diet been unsatisfactory because of problems with your teeth of mouth? Have you had to interrupt meals because of problems with your teeth or mouth? Have you found it difficult to relax because of problems with your teeth or mouth? Have you been a bit embarrassed because of problems with your teeth or mouth? Have you been a bit
Attached mucosa measurement | 0 day
  The width of the keratinised attached mucosa is measured using the UNC-15 periodontal probe. This is done by determining the mucosa-gingival junction line on the vestibular side. The distance from this line to the apex of the alveolar ridge will correspond to the width of the keratinised attached mucosa.
Attached mucosa measurement | 90 days
  The width of the keratinised attached mucosa is measured using the UNC-15 periodontal probe. This is done by determining the mucosa-gingival junction line on the vestibular side. The distance from this line to the apex of the alveolar ridge will correspond to the width of the keratinised attached mucosa.

CONTACTS AND LOCATIONS:
Locations (1):
- I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
IPD Sharing is impossible because of the recommendation of the local ethics committee